CLINICAL TRIAL: NCT05354726
Title: Investigation of Skeletal and Respiratory Muscle Strength, Pulmonary Function, Exercise Capacity and Physical Activity in Children With Chronic Kidney Disease
Brief Title: Skeletal and Respiratory Muscle Strength, Pulmonary Function, Exercise Capacity and Physical Activity in Pediatric Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Haluk TEKERLEK, Principal Investigator/Research Assistant, Hacettepe University
Other Study IDs: pedichronickidneydisease
Record Dates: First submitted 2022-04-20; First posted 2022-04-29 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CKD group: Inclusion Criteria for Volunteers (Inclusion Criteria):
  * 6-18 age range,
  * According to the Chronic Kidney Disease Assessment and Classification Guide prepared by the National Kidney Foundation- Kidney Disease Outcomes Quality Initiative (NKF-KDOQI); Stage 2, glomerular filtration rate 60-89 ml/min/1.73 m2, Stage 3, glomerular filtration rate 30-59 ml/min/1.73 m2, Stage 4, glomerular filtration rate 15-29 ml/min/1.73 m2,
  * Presence of kidney transplantation was determined as inclusion criteria.
  Exclusion Criteria for Volunteers:
  * acute infection,
  * Ongoing dialysis,
  * Congenital heart disease,
  * Hypertension that cannot be controlled with dual antihypertensive medication,
  * Neurological and/or genetic musculoskeletal disease,
  * The presence of orthopedic and cognitive problems that prevented the tests from being performed were determined as exclusion criteria.
  Interventions: Other: Assessments parameters
- Control Group: Inclusion Criteria for Control Volunteers:
  * Not have cardiovascular, neurological and/or genetic musculoskeletal disease
  * Not having orthopedic and cognitive problems that prevent testing
  * The patient's and/or family's willingness to participate in the study
  Interventions: Other: Assessments parameters

INTERVENTIONS:
Other: Assessments parameters — Demographic and Clinical Characteristics, Bone Mineral Density, Sarcopenia, Body Composition, Arterial Stiffness, Endothelial Function, Echocardiography,Pulmonary Function, Respiratory Muscle Strength, Submaximal exercise capacity, Maximal Exercise Capacity, Physical Activity Level, Hand Grip Strength, Lower Extremity Muscle Strength

SUMMARY:
Studies examining musculoskeletal strength, respiratory function and muscle strength, physical activity level and exercise capacity in children with CKD and evaluating the relationships between these parameters have not been found both in the world and in our country. In this study, it is aimed to evaluate skeletal and respiratory muscle strength, respiratory parameters and exercise capacity in children with CKD primarily and compare them with healthy children. Secondly, it is to examine the relationship between endothelial function, arterial stiffness, sarcopenia and physical activity in children with CKD. It is thought that the results to be obtained with the study will support the literature with the prediction that rehabilitation programs for patients in all stages of CKD will be structured and in this way will contribute positively to the management and prognosis of the disease.

Hypotheses H0: There is no difference between children with chronic kidney disease and healthy children in terms of skeletal and respiratory muscle strength, respiratory parameters and exercise capacity.

H1: There is a difference between children with chronic kidney disease and healthy children in terms of skeletal and respiratory muscle strength, parameters and exercise capacity.

H0: There is no relationship between endothelial function, arterial stiffness, sarcopenia and physical activity in children with chronic kidney disease.

H1: There is a relationship between endothelial function, arterial stiffness, sarcopenia and physical activity in children with chronic kidney disease.

DETAILED DESCRIPTION:
Children who applied to Gazi University, Faculty of Medicine, Department of Pediatrics, Department of Pediatric Nephrology and met the specified inclusion criteria will be included in our study. Patients will be referred to Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit after the routine evaluations including demographic and clinical characteristics, laboratory tests and anthropometric measurements are completed. Here, patients will be evaluated with physical therapy and rehabilitation measurement and evaluation methods such as muscle strength, exercise capacity and physical activity. The healthy control group will be formed by inviting the healthy relatives of the patients who applied to our faculty to participate in the study. After obtaining informed consent, healthy children will be evaluated.

Details of Working Method For each child with chronic kidney disease, age, gender, body weight, height, systolic and diastolic blood pressure, and results of routine blood tests (complete blood count test parameters: hemoglobin, hematocrit, erythrocyte, leukocyte and platelet count) biochemistry test parameters (blood sugar, blood urea nitrogen, creatinine, uric acid, sodium, potassium, chlorine, calcium, phosphorus, alkaline phosphatase, total protein, albumin, alanine aminotransferase, aspartate aminotransferase, triglyceride, total cholesterol, high-density lipoprotein, low-density lipoprotein levels , venous blood pH and bicarbonate etc. values), ferritin, parathormone, 25 hydroxy vitamin D level) will be recorded. The age at diagnosis, duration and etiology of the disease, current treatment information and drugs used will be recorded. Body composition data will also be recorded for children with CKD. Bone mineral density parameters in the last six months, left ventricular mass index values in the last three months, 24-hour blood pressure monitoring (ABPM) in the last month, and heart rate measured on the same device are used in the follow-up of the patients. wave velocity (pulse wave velocity-PWV) evaluation results will be used, if there is none, ABPM and PWV will be performed again. After these evaluations, parameters such as skeletal muscle strength, respiratory muscle strength, and exercise capacity will be evaluated in both the patient group and healthy children, and the obtained data will be compared. In addition, the relationship between parameters such as complete blood count parameters, biochemistry test parameters, routine bone markers, BMD, heart and vascular function evaluations and parameters such as skeletal and respiratory muscle strength, exercise capacity, and physical activity level will be examined in children with CKD. In case of adequate data, children with CKD will be subgrouped according to disease stage and assessment data will be analyzed by subgroups.

ELIGIBILITY:
Group: CKD group

Inclusion Criteria for Volunteers (Inclusion Criteria):

* 6-18 age range,
* According to the Chronic Kidney Disease Assessment and Classification Guide prepared by the National Kidney Foundation- Kidney Disease Outcomes Quality Initiative (NKF-KDOQI); Stage 2, glomerular filtration rate 60-89 ml/min/1.73 m2, Stage 3, glomerular filtration rate 30-59 ml/min/1.73 m2, Stage 4, glomerular filtration rate 15-29 ml/min/1.73 m2,
* Presence of kidney transplantation was determined as inclusion criteria.

Exclusion Criteria for Volunteers:

* acute infection,
* Ongoing dialysis,
* Congenital heart disease,
* Hypertension that cannot be controlled with dual antihypertensive medication,
* Neurological and/or genetic musculoskeletal disease,
* The presence of orthopedic and cognitive problems that prevented the tests from being performed were determined as exclusion criteria.

Group: Control Group

Inclusion Criteria for Control Volunteers:

* Not have cardiovascular, neurological and/or genetic musculoskeletal disease
* Not having orthopedic and cognitive problems that prevent testing
* The patient's and/or family's willingness to participate in the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children who applied to Gazi University, Faculty of Medicine, Department of Pediatrics, Department of Pediatric Nephrology and met the specified inclusion criteria will be included in our study. Patients will be referred to Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit after the routine evaluations including demographic and clinical characteristics, laboratory tests and anthropometric measurements are completed. Here, patients will be evaluated with physical therapy and rehabilitation measurement and evaluation methods such as muscle strength, exercise capacity and physical activity. The healthy control group will be formed by inviting the healthy relatives of the patients who applied to our faculty to participate in the study. After obtaining informed consent, healthy children will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
Bone mineral density (BMD) z-score | 15-25 minutes
  Bone mineral density (BMD) measurement will be measured with a double X-ray absorptiometry device (DEXA (Horizon Wi (S/N 300796M))). Lumbar vertebral total BMD value and BMD z score will be calculated for each child. BMD z score -1 standard between -2 and -2 standard deviations, it will be considered as osteopenia, if it is less than -2 standard deviations, it will be considered as osteoporosis.This evaluation parameter will be recorded from the most recent test results for diagnosis and clinical course.
Skeletal muscle mass (SMM) z-score | 15-25 minutes
  Total/regional (obsolute/t-score and z-score) fat mass, lean mass (lean mass) and lean-boneless mass (lean mass) will be measured by dual energy X-ray absorptiometry device (DEXA (device tag). Skeletal muscle mass ( SMM), SMM z score and appendicular lean-boneless mass (appendicular lean mass) will be calculated according to the SMM values of healthy children based on age and gender.If the SMM z score is below -2 standard deviations, it will be considered as sarcopenia.
Arterial stiffness | 10 minutes
  Arterial stiffness will be assessed using the pulse wave velocity (PWV) technique with the blood pressure holter-ABPM (spacelabs) device. Pulse waves will be recorded by placing the proximal sensor of the device in the places where the carotid artery and the distal sensor of the femoral artery are best palpated. The distance between these two points and the pulse propagation velocity will be calculated with the help of a computer in m/sec. High velocity data indicates high arterial stiffness, low velocity indicates less arterial stiffness.
Carotid artery intima-media thickness (cIMT) | 10-15 minutes
  For endothelial function, standardized measurement of carotid artery intima-media thickness (cIMT) will be made by the same radiologist with a high-resolution US device (General Electric) with a multi-frequency liner probe (5-12 MHz). Measurements will be taken over the bilateral distal common carotid arteries (1 cm proximal to bufircation) while the patients are supine and their necks are in neutral extension. cIMT is defined as the distance between the lumen-intima interface and the media-adventitia interface. A total of 6 records, three from each side, will be taken and the average will be recorded as cIMT.
Left ventricular mass index | 10-15 minutes
  Left ventricular mass index measurement and evaluation of left ventricular hypertrophy will be performed. Interventricular septum, posterior wall and left ventricular wall thickness measurements will be taken in diastole with M mode echocardiography. The presence of LVH will be evaluated by evaluating the left ventricular mass (LVMI) calculated and indexed by using the Devereux formula according to age, gender and height.
Forced expiratory volume in 1 second (FEV1) | 10-15 minutes
  Pulmonary function testing will be performed with a portable spirometer (Spirodoc, Medical International Research, Rome, Italy) using standard procedures. Forced expiratory volume in 1 second (FEV1), will be saved.
Forced vital capacity (FVC) | 10-15 minutes
  Pulmonary function testing will be performed with a portable spirometer (Spirodoc, Medical International Research, Rome, Italy) using standard procedures. Forced vital capacity (FVC) parameter will be saved.
FEV1/FVC | 10-15 minutes
  Pulmonary function testing will be performed with a portable spirometer (Spirodoc, Medical International Research, Rome, Italy) using standard procedures. FEV1/FVC parameter will be saved.
Maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) | 10-15 minutes
  Maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) will be used as indicators of respiratory muscle strength (28). A portable intraoral pressure gauge (MicroRPM, Micromedical, Kent, UK) and nose clip will be used during MIP and MEP assessments. MIP and MEP measurements will be obtained using standard procedures. 3 measurements will be made where the difference between each measurement is not more than 10% and the maximum value of MIP and MEP will be recorded.
6-Minute Walk Test (6 MWT) distance | 10-15 minutes
  Submaximal exercise capacity will be evaluated with the 6-Minute Walk Test (6 MWT). The standard protocol will be implemented in a continuous corridor of 30 meters. The patient wearing comfortable clothes and shoes will be given standard instructions and verbal guidance during the test. The distance the patient walked during the test will be recorded in meters.
ISWT distance | 10-15 minutes
  Maximal exercise capacity will be evaluated with the incremental shuttle walk test (ISWT). For the ISWT, it will be adjusted to a total of 10 meters with 2 cones placed at a distance of 9.0 meters from each other and a rotational margin of 0.5 meters. In this system, the patient will be asked to walk in a round-trip way, adapting to the increasing speed and the sound coming from outside. In the shuttles that are getting faster and faster, the lap number of the patients, the number of laps of the last level they can reach, and the walking/running distances in meters will be recorded.
Physical Activity Level | 5-10 minutes
  The scale to be used for this purpose is the Child Physical Activity Questionnaire (MFAA) developed by Kowalski et al. It is a seven-day self-reported recall scale designed to assess moderate-intensity physical activity in children aged 8-14 years. CFAA is designed to be implemented throughout the school year. The Turkish validity and reliability of the questionnaire was made and permission was obtained from the responsible author for its use.
Hand Grip Strenght | 10-15 minutes
  Hand grip strength will be measured using a hand dynamometer (Jamar, Sammons Preston, Rolyon, Bolingbrook, IL). Measurements will be made using standard procedures, right and left sides, with the arms at the side of the trunk, the elbow in a 90-degree flexion position, and the forearm and wrist in a neutral position. The highest of the three measurements will be considered as hand grip strength.
Maximum isometric muscle strength of the quadriceps femoris | 10-15 minutes
  Maximum isometric muscle strength of the quadriceps femoris muscle will be measured with a dynamometer (Lafayette Instrument Company, Lafayette, Indiana).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University and Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided